CLINICAL TRIAL: NCT05234307
Title: A Phase Ib Trial of PBF-1129 and Nivolumab in Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: PBF-1129 and Nivolumab for the Treatment of Recurrent or Metastatic Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dwight Owen (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Dwight Owen, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-21156; NCI-2022-00236 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R01CA248741 (NIH)
Record Dates: First submitted 2022-02-01; First posted 2022-02-10 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Lung Non-Small Cell Carcinoma; Recurrent Lung Non-Small Cell Carcinoma; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (PBF-1129, nivolumab) (Experimental): Patients receive PBF-1129 PO QD and nivolumab IV on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Adenosine A2B Receptor Antagonist PBF-1129; Procedure: Biospecimen Collection; Biological: Nivolumab

INTERVENTIONS:
Drug: Adenosine A2B Receptor Antagonist PBF-1129 — Given PO
  Other Names: A2BR Antagonist PBF-1129; PBF 1129; PBF-1129; PBF1129
Procedure: Biospecimen Collection — Correlative studies
  Other Names: Biological Sample Collection; Biospecimen Collected
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; CMAB819; MDX-1106; NIVO; Nivolumab Biosimilar CMAB819; ONO-4538; Opdivo

SUMMARY:
This phase I trial studies the side effects and best dose of PBF-1129 in combination with nivolumab in treating patients with non-small cell lung cancer that has come back (recurrent) or spread to other places in the body (metastatic). Immunotherapy with monoclonal antibodies, such as PBF-1129 and nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety and tolerability of the combination of adenosine A2B receptor antagonist PBF-1129 (PBF-1129) and nivolumab in patients with advanced non-small cell lung cancer (NSCLC) based upon the Common Terminology Criteria for Adverse Events (CTCAE) version 5 criteria.

SECONDARY OBJECTIVE:

I. To determine the efficacy of the combination of PBF-1129 and nivolumab in patients with advanced NSCLC, including progression-free survival (PFS), objective response (ORR), disease control rate (DCR), and overall survival (OS) based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

EXPLORATORY OBJECTIVES:

I. To study the effect of PBF-1129 on the levels of myeloid-derived suppressor cells (MDSC) within the tumor microenvironment (TME) and in peripheral blood of study patients.

II. To evaluate correlative biomarkers that might predict disease response to treatment with PBF-1129 and nivolumab therapy in previously treated NSCLC patients including STK11 genetic alterations and a transcriptional signature of LKB1 functional status developed by the Carbone lab.

OUTLINE: This is a dose-escalation study of PBF-1129 given in combination with immune checkpoint blockade.

Patients receive adenosine A2B receptor antagonist PBF-1129 (PBF-1129) orally (PO) once daily (QD) and nivolumab intravenously (IV) on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 12 weeks for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Confirmed recurrent or metastatic non-small cell carcinoma of the lung of any histology without curative options
* Measurable disease based on RECIST 1.1
* Patients must have received standard of care chemotherapy and immunotherapy. No limits to prior lines of therapy. Prior PD-1 and/or PD-L1 directed therapies are required. Prior CTLA4 therapy is permitted. Patients may have received no more than 3 prior lines of therapy in the metastatic setting (excluding targeted therapies)
* Patients with known actionable mutations with Food and Drug Administration (FDA)-approved treatment options must have received all approved and standard of care treatment options (ie osimertinib for EGFR, alectinib for ALK, etc)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Absolute neutrophil count (ANC) >= 1,500 /mcL
* Platelets >= 100,000 / mcL
* Serum creatinine OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) =< 1.5 X upper limit of normal (ULN) OR >= 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN
* Serum total bilirubin =< 1.5 X ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN
* AAspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 X ULN OR =< 5 X ULN for subjects with liver metastases
* Albumin >= 2.5 mg/dL
* International normalized ratio (INR) or prothrombin time (PT) or activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Anticipated life expectancy of >= 3 months
* Willing to comply with study procedures
* Must be able to swallow pills
* Female subjects of childbearing potential must be willing to use an adequate method of contraception
* For female patients of childbearing potential, a negative serum pregnancy test within 7 days prior to first dose of protocol therapy is required
* Be willing and able to understand and sign the written informed consent document
* Availability of a recent formalin-fixed, paraffin-embedded (FFPE) tumor tissue block. A recently obtained archival FFPE tumor tissue block (if an FFPE tissue block cannot be provided, 15 unstained slides (10 minimum) will be acceptable) from a primary or metastatic tumor resection or biopsy can be provided if it was obtained within 1 year of trial screening. Patients with archival tissue that does not meet this criteria may still be eligible in the dose escalation cohort only upon approval from PI.
* For patients in dose expansion cohort: Be willing to provide tissue from a pre-treatment and on-treatment fin needle aspirate (FNA) or core biopsy of a tumor lesion. Subjects must consent to pre-treatment and on-treatment biopsy prior to initiation of clinical trial, however subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may still continue on study
* Be willing to provide peripheral blood samples for correlative studies

Exclusion Criteria:

* Has active autoimmune disease, including myasthenic syndrome, which has required systemic treatment in the past 12 months (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided that disease is well controlled at baseline and requires only topical corticosteroids.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (at a dose > 10 mg prednisone or equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Known active chronic infections - human immunodeficiency virus (HIV)/acquired immunodeficiency syndrome (AIDS), known active (ie with detectable polymerase chain reaction [PCR]) Hepatitis B or C
* Cirrhosis (Child-Pugh B or worse) or cirrhosis with history of hepatic encephalopathy or clinically meaningful ascites resulting from cirrhosis. Clinically meaningful ascites is defined as ascites from cirrhosis requiring diuretics or paracentesis
* Symptomatic central nervous system (CNS) metastases. Patients with treated brain metastases are eligible if they are clinically stable with regard to neurologic function, on stable dose of steroids after cranial irradiation with maximum of 10 mg prednisone equivalent. Treatment (whole brain radiation therapy, focal radiation therapy, and stereotactic radiosurgery) must be completed at least 2 weeks prior to study entry, or after surgical resection performed at least 28 days prior to treatment initiation. Patients with asymptomatic lesions will be eligible if considered appropriate by the treating physician.
* Pregnancy or breastfeeding
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Any of the following cardiac criteria:

  * Mean resting corrected QT interval (corrected QT [QTc] using Fredericia's formula [QTcF]) > 470 msec (Fridericia's Criteria for Corrected QT interval [QTc] Calculation: Fridericia's formula QTcF = (QT/RR0.33). RR is the time from the interval of 1 QRS complex to the next measured in seconds and is commonly calculated as (60/heart rate [HR])
  * Any clinically important abnormalities in rhythm, conduction or morphology of resting electrocardiogram (ECG) (e.g., complete left bundle branch block, third degree heart block, second degree heart block
* Any patient who experience unacceptable toxicity on prior checkpoint inhibitor therapy:

  * >= grade 3 adverse event (AE) related to checkpoint inhibitor with the exception of grade 3 pneumonitis that has resolved to grade 1 at time of study entry.
  * Ongoing >= grade 2 immune-related AE associated with checkpoint inhibitor with the exception of endocrine toxicities as detailed below
  * CNS, ocular or cardiac AE of any grade related to checkpoint inhibitor
  * NOTE: Patients with a prior endocrine AE are permitted to enroll if they are stably maintained on appropriate replacement therapy and are asymptomatic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 30 days after the last dose of study treatment
  Safety will be measured by the occurrence of dose-limited toxicities as well as any other adverse events as defined in Common Terminology Criteria for Adverse Events version 5. Frequency and severity of adverse events and tolerability of the regimen will be collected and summarized by descriptive statistics. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns. All patients who have received at least one dose of the therapeutic agents will be evaluable for toxicity and tolerability.

SECONDARY OUTCOMES:
Overall objective response rate | Up to 1 year after treatment discontinuation
  Will be calculated and exact binomial 95% confidence interval (CI) will be provided.
Disease control rate | Up to 1 year after treatment discontinuation
  Will be calculated and exact binomial 95% CI will be provided.
Overall survival | Up to 1 year after treatment discontinuation
  Will be defined as time from initiation of therapy to death, or censored at last follow-up date if the subject is alive. Kaplan-Meier methods will be used to estimate overall survival with 95% CI.
Progression free survival | Up to 1 year after treatment discontinuation
  Will be defined as the time from initiation of therapy to the time of Response Evaluation Criteria in Solid Tumors progression or death. Kaplan-Meier methods will be used to estimate progression free survival with 95% CI.

OTHER OUTCOMES:
Levels of myeloidderived suppressor cells (MDSC) | Up to 1 year after treatment discontinuation
  Baseline MDSC and the changes upon treatment will be compared between responders and non-responders using two sample t-test or non-parametric Wilcoxon test as appropriate. Linear mixed effect models will be used to evaluate MDSC levels over the time with the response, as well as the clinical outcomes including resistance to treatment. Potential confounders (patients' demographics and clinical characteristics) might be included in the models.
Correlative biomarkers | Up to 1 year after treatment discontinuation
  We will compare responses within this cohort. The impact of STK11/LKB1 alterations and how it is associated with response will be assessed using logistic regression analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Dwight H Owen, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu